CLINICAL TRIAL: NCT07225101
Title: Evaluation of the Efficacy of STRATAFIX for Neurosurgical Cranial and Spine Procedures
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Michael Karsy, Assistant Clinical Professor of Neurosurgery, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00268953
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Wound Closure; Brain Tumor Adult; Spine; Neurovascular; Hemorrhagic Stroke, Intracerebral; Traumatic Brain Injury
Keywords: Superficial surgical site infection; Suture material; Wound closure techniques; brain tumor; spine; spine trauma; neurosurgery; hemorrhagic stroke; traumatic brain injury
MeSH Terms: conditions — Hemorrhagic Stroke; Brain Injuries, Traumatic; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label, single-arm, non-crossover prospective cohort study with non-inferiority statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- STRATAFIX PDS and Monocryl suture (Experimental): All participants enrolled will have their scheduled surgery as planned with their wound closed using STRATAFIX.
  Interventions: Device: STRATAFIX PDS and Monocryl suture

INTERVENTIONS:
Device: STRATAFIX PDS and Monocryl suture — STRATAFIX, suture employs a novel incorporation of barbed components to suture resulting in tension holding closure with long-lasting absorbable suture.

SUMMARY:
This research is studying a device already approved by the Food and Drug Administration (FDA) to treat wound closures. Researchers are studying a large group of people to continue to learn information about the safety of the STRATAFIX suture and how people's bodies react to using it over a long period of time. This research will provide additional information about using STRATAFIX sutures to close surgical wounds.

ELIGIBILITY:
Inclusion Criteria:

* Elective or emergent surgical approaches for cranial or spine neurosurgical approaches, requiring sutures for wound closure, requiring multilayer wound closure

Exclusion Criteria:

* Patients with prior surgical wound dehiscence or infection
* Patients with allergy to suture material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound complications Bates-Jensen Wound Assessment Tool (BWAT) score | 1 month
  The BWAT evaluates 13 categories including size, depth, edges, undermining, necrotic tissue type and amount, exudate type and amount, skin color, peripheral tissue, granulation tissue and epithelialization with a total score of 65. Minimal severity scores are 10-20 out of the total of 65 with good interrater reliability and validation in a variety of clinical environments. Wounds with scores <10 will be considered healed.

SECONDARY OUTCOMES:
Wound complications Bates-Jensen Wound Assessment Tool (BWAT) score | 3 and 6 months
  The BWAT evaluates 13 categories including size, depth, edges, undermining, necrotic tissue type and amount, exudate type and amount, skin color, peripheral tissue, granulation tissue and epithelialization with a total score of 65. Minimal severity scores are 10-20 out of the total of 65 with good interrater reliability and validation in a variety of clinical environments. Wounds with scores <10 will be considered healed.
  Scores will be separated into specific patient subgroups (e.g., spine procedures vs. cranial procedures, younger vs. older patients)
The Wound-Quality of Life (QOL) questionnaire score | 1, 3 and 6 months
  This is a 17-point scale with 5 choices each ranging from 17-85. Higher scores indicate worse quality of life.
Intraoperative time required for wound closure | Immediately following surgery
  Time for intraoperative wound closure will be monitored. Wound closure technique will be video recorded.
Percent of participants positive for superficial surgical site infection (SSI) | Up to six months
  Assessed using a culture or polymerase chain reaction
Number of case deviations and descriptions from prescribed suturing paradigm | Immediately following surgery
  A quantification and description for additional suture material required for surgical procedures will be monitored.
Liker scale of patient satisfaction with wound | 1, 3 and 6 months
  10 point subjective scale indicating patient satisfaction with wound
Wound imaging at perioperative followup | 1, 3 and 6 months
  Wound pictures during followup period.
Wound revision strategy | up to 6 months
  Description of any wound revision strategies and timing

CONTACTS AND LOCATIONS:
Overall Officials: Michael Karsy, MD, PhD, MSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health Sparrow, Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
Unclear if manuscript will be published in an ICMJE journal and data from this study are restricted from the University of Michigan Data Use Committee